CLINICAL TRIAL: NCT02229916
Title: Swiss Austrian German Testicular Cancer Cohort Study - SAG TCCS
Acronym: SAG TCCS
Status: Recruiting | Type: Observational
Sponsor: Dr. med. Christian Rothermundt (Other)
Collaborators: German Testicular Cancer Study Group (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Christian Rothermundt, PD Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: SG359/13
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Testicular Neoplasms
Keywords: Testicular Neoplasms; Testicular Cancer; Cohort Study
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The majority of testicular cancer patients can be cured with cisplatin-based chemotherapy. Mortality has been reduced even more within the last 15 years due to the stringent application of standard chemotherapy followed by resection of residual disease. This is a positive development considering that testicular cancer usually affects young men. Active surveillance has become an acceptable and widely used strategy in stage I testicular cancer. Thus, it is important to follow these patients in a standardized way and to adhere to a rationale surveillance strategy. There is no international consensus regarding follow-up of testicular cancer patients. Stratification according to risks and patterns of relapse would allow to tailor follow-up schedules, aiming at early identification of relapse without causing unnecessary harm by using excessive radiation in these young long-term survivors. Follow-up procedures should not only aim at detecting relapse, but also long-term side effects from therapy, including hypogonadism, metabolic syndrome, cardiovascular disease and secondary malignancies. The Swiss Austrian German Testicular Cancer Cohort Study (SAG TCCS) will comprise consecutive newly diagnosed testicular cancer patients and is the first study to prospectively evaluate the initial indictor of relapse in testicular cancer patients, the frequency and pattern of relapse and document long-term toxicities of the treatment (cardiovascular, gonadal, hearing impairment, renal function and second malignancies) and psychosocial aspects. This cohort study will determine the relevance of each test performed routinely during follow-up. The collected data will have direct implications for the care of patients with testicular cancer and inform future adaptations of follow-up recommendations. The dataset will give information on baseline factors of testicular cancer patients patients, current treatment strategies in Switzerland, Austria and Germany, outcome and late sequelae.

DETAILED DESCRIPTION:
Objectives

Primary objective

The primary objective is to determine the diagnostic performance and the clinical impact of a variety of tests, including conventional radiographs, computer tomographies (CT), abdominal ultrasound, serum tumour markers (AFP, beta-HCG and LDH) and clinical signs and symptoms aimed at early detection of relapse after curative therapy with documented complete remission.

Secondary objectives

Diagnostic performance:

1. To determine the rate of relapses detected on chest x-ray in seminoma patients.
2. To determine the rate of false positive abnormalities on CT scan and of false positive tumour marker elevations not due to seminomatous or non-seminomatous germ cell tumour relapses but due to other processes.
3. To determine the modality to rule out testicular cancer relapse in patients with false positive index tests.

   Pattern of care:
4. To assess patient characteristics at baseline and at the time-point of relapse detection.
5. To determine the rate of stage I seminoma and non-seminoma patients undergoing active surveillance.
6. To obtain an overview of treatment and follow-up strategies in germ cell cancer patients in Switzerland.

   Outcome:
7. To collect data on treatment sequelae following testicular cancer treatment in terms of organ function, cardiovascular risk factors, sexual health and socioeconomic aspects.
8. To determine the rate of intermediate and poor-prognosis disease at relapse.
9. To determine the rate of offspring spontaneously conceived after testicular cancer treatment.

Design

Prospective cohort study

Centres All urologists, radiooncologists and oncologists are motivated to enrol their patients. We will aim at enrolling the majority of patients treated and followed in private practice.

Patients Consecutive patients with testicular cancer of any type and any stage (incident cases). Testicular cancers are generally classified as seminomatous (seminoma) and nonseminomatous germ cell tumours (non-seminoma) of the testis. Mixed germ cell tumours belong to the group of non-seminomas. The stage of disease and the choice of treatment (active surveillance vs. chemotherapy vs. radiotherapy) define the risk of relapse, the pattern of relapse and the long-term toxicities. Staging in testicular cancer is performed according to the American Joint Committee on Cancer (AJCC) primary tumor, regional nodes, metastasis (TNM) staging system for testis cancer. Metastatic testicular cancers are classified according to the International Germ Cell Cancer Collaborative Group (IGCCCG) risk groups.

Clinical outcome

Relapse of testicular cancer will be defined as rising concentrations of serum alphafetoprotein (AFP) above the upper limit of normal (typically > 13 μg/l) and/or human chorionic gonadotropin (HCG) above the upper limit of normal (typically > 5 U/l) and/or lactate dehydrogenase (LDH) above the upper limit of normal and confirmation of this rise in a second test four weeks later and/or radiographic evidence of metastatic disease in typical locations, and/or the presence of active germ cell tumour established by biopsy, whatever comes first.

Index tests

The following tests will be performed (ordered according to their burden for patients and cost): symptom assessment, physical examination, tumour marker measurement, chest x-ray, abdominal ultrasound and CT scan of abdomen and pelvis.

Procedures

Follow-up will be performed according to the mandatory follow-up schedule by a physician who has substantial experience in the treatment and surveillance of patients with germ cell tumours. Follow-up comprises thorough assessment of medical history and patients' symptoms with a focus on pain, appetite, fatigue, sexual function and activities of daily living; physical examination includes lung auscultation, abdominal, axillary, supra- and infradiaphragmatic regional lymph nodes and testicular palpation; serum tumour marker measurement: AFP, HCG and LDH; chest x-ray and abdominal ultrasound or CT scan. Even though the role of LDH in the follow-up is debatable, due to limited sensitivity and specificity and a high rate of false-positive tests, it can contribute to identify relapse in a significant number of cases, as shown in a recent publication. All the laboratory and radiological tests are performed independently and results are not made available to the investigator prior to symptom assessment and physical examination. In addition we will ascertain cardiovascular risk factors (smoking status, lipid profile, bodymass index, fasting glucose etc.), renal function, testosterone level, follicle stimulating hormone (FSH) level, lutenizing hormone (LH) level, and socioeconomic characteristics (education, employment, partnership) in annual intervals.

Statistics

Sample size considerations

There are approximately 400 newly diagnosed testicular cancer patients in Switzerland per year. In Germany the annual testicular cancer incidence is about 4000. We aim at including approximately 300 patients per year in Switzerland over a duration of 3 years, with a total number of 900 patients. We are also aiming at registration of 2000 patients per year in Germany. Looking at the Swiss cohort, with an estimated 15% rate of relapses over a follow-up duration of two years, this will yield approximately 135 cases with relapse. This number will yield satisfactory statistical precision. An assumed sensitivity of 50% and a specificity of 95% for Beta-HCG, for example, to detect a relapse will yield a positive likelihood ratio (LR) of 10 and a negative likelihood ratio of 0.53. Corresponding 95% confidence intervals will be 42 to 58% for sensitivity, 93 to 97% for specificity, 7.0 to 14.2 for the positive likelihood ratio and 0.44 to 0.62 for the negative likelihood ratio. An assumed sensitivity of 37% and a specificity of 99% for CT scans, for example, to detect a relapse will yield a positive likelihood ratio of 37 and a negative likelihood ratio of 0.64. Corresponding 95% confidence intervals will be 29 to 45% for sensitivity, 98 to 100% for specificity, 17.7 to 77.4 for the positive likelihood ratio and 0.56 to 0.72 for the negative likelihood ratio.

Measures of diagnostic accuracy will be determined in relation to the occurrence and timepoint of diagnosis of a relapse as specified above. Tests that were positive within the previous 8 weeks of established diagnosis of relapse will be considered as true positives, tests that remained negative during this time period as false negatives. Conversely, tests that were positive before this time period will be considered as false positives, and tests that were negative before this period as true negatives. We will use a multi-level model with random effects at the level of patients and time-points to estimate sensitivities and specificities and likelihood ratios, with the data organised in long format, with each test outcome (positive or negative) at each time-point represented by one line in the dataset, determining for each time-point whether it is within the 8-week time-period previous to the time-point of established diagnosis of relapse. The model takes into account the correlation of multiple time-points and tests within patients. The positive LR indicates how much more likely it is to find a positive test in patients with a relapse (sensitivity) as compared with those without relapse (1-specificity). Conversely, the negative LR specifies how much less likely it is to find a negative test in patients with relapse (1-sensitivity) as compared to patients without (specificity). A test will be considered to provide clinically relevant power to rule in or out a relapse if the positive and negative LRs are above 5 or below 0.2, respectively. The test will be considered to have a strong power to rule in or out a relapse if LRs are above 10 or below 0.1, respectively.

As measures of the clinical impact of the addition of more extensive tests, we will examine the net re-classification improvement and the integrated discrimination improvement. The net re-classification improvement through the addition of a more extensive test is defined as the improvement of the probability of the appropriate classification of patients according to relapse status (presence or absence of a relapse), which is afforded by the addition of the more extensive test. This corresponds to the sum of differences in proportions of individuals classified positive minus the proportion classified negative for individuals who develop events, and the proportion of individuals classified negative minus the proportion classified positive for individuals who do not develop events. The integrated discrimination improvement is defined as the improvement in average sensitivity afforded by the addition of the more extensive test minus the potential loss in specificity afforded by the addition of the more extensive test. All analyses will be done using Stata, Release 11 (Stata Corp LP, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histologically proven seminomas or non-seminoma.
* Seminoma: complete remission (CR) or lymph nodes (LN) < 3cm or PET negative partial remission (PR) or non-seminoma: CR.
* Completion of treatment within the last 6 months.
* Patient able and willing to attend for regular surveillance.

Exclusion Criteria:

* Co-existent malignancy within 5 years.
* Inability for any reason to comply with the trial investigations or follow-up schedules.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with testicular cancer of any type and any stage and any age (incident cases).
  Testicular cancers are generally classified as seminomatous (seminoma) and nonseminomatous germ cell tumours (nonseminoma) of the testis. Mixed germ cell tumours belong to the group of non-seminomas. The stage of disease and the choice of treatment (active surveillance vs. chemotherapy vs. radiotherapy) define the risk of relapse, the pattern of relapse and the long-term toxicities. Staging in testicular cancer is performed according to the American Joint Committee on Cancer (AJCC) TNM staging system for testis cancer [46]. Metastatic testicular cancers are classified according to the International Germ Cell Cancer Collaborative Group (IGCCCG) risk groups [47].
Sampling Method: Non-Probability Sample
Enrollment: 6900 (Estimated)
Dates: Start 2013-12; Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Mode of relapse detection | 8 years
  Diagnostic performance and the clinical impact of a variety of tests, including conventional radiographs, computed tomographies (CT), abdominal ultrasound, serum tumour markers (AFP, beta-HCG and LDH) and clinical signs and symptoms aimed at early detection of relapse after curative therapy with documented complete remission.

SECONDARY OUTCOMES:
Rate of relapses detected on chest x-ray in seminoma patients | 8 years
Rate of false positive abnormalities on CT scan | 8 years
Rate of false positive tumour marker elevations not due to seminomatous or non-seminomatous germ cell tumour relapses but due to other reasons | 8 years
Patient characteristics at baseline and at the time-point of relapse detection. | 8 years
Rate of stage I seminoma and non-seminoma patients undergoing active surveillance. | 8 years
Overview of treatment and follow-up strategies in germ cell cancer patients in Switzerland, Austria and Germany | 8 years
Treatment sequelae following testicular cancer treatment in terms of organ function, cardiovascular risk factors, sexual health and socioeconomic aspects. | 8 years
Rate of intermediate and poor-prognosis disease at relapse. | 8 years
Rate of offspring spontaneously conceived after testicular cancer treatment. | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rothermundt, Dr. med., Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Kantonsspital St.Gallen; Onkologie/Haematologie, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] Rothermundt C, Thurneysen C, Cathomas R, Muller B, Mingrone W, Hirschi-Blickenstorfer A, Wehrhahn T, Ruf C, Rothschild S, Seifert B, Terbuch A, Grassmugg T, Woelky R, Fankhauser C, Kunit T, Fischer N, Inauen R, Kamradt J, Ziegler K, Haynes A, Juni P, Gillessen S. Baseline characteristics and patterns of care in testicular cancer patients: first data from the Swiss Austrian German Testicular Cancer Cohort Study (SAG TCCS). Swiss Med Wkly. 2018 Jul 24;148:w14640. doi: 10.4414/smw.2018.14640. eCollection 2018. PMID 30044478
- See also: Webpage with basic information on the cohort study and link to the electronic case report form (eCRF) portal — http://www.sag-tccs.com/